CLINICAL TRIAL: NCT04715685
Title: Mind Body Balance for Pediatric Migraine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MOST Study; U01AT010132 (NIH)
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Headache; Headache Disorders; Headache, Migraine; Migraine; Migraine Disorders; Migraine With Aura; Migraine Without Aura; Chronic Migraine
Keywords: headache; migraine; cognitive behavioral therapy; pediatrics; mind body intervention; diaphragmatic breathing; progressive muscle relaxation; imagery; relaxation; biofeedback
MeSH Terms: conditions — Headache; Headache Disorders; Migraine Disorders; Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only than study staff whose role requires unblinding (project manager and the nurse or interventionist providing the treatment) will be made aware of each participant's study assignment by the statistician. Other study personnel (including assessors of key variables) will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 40 minute session, home practice e-health, phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 40 minutes in duration. The daily home practice component for headache management will utilize a migraine specific interactive web portal, Migraine e-health portal. This arm will also receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 40 minute session; Behavioral: home practice e-health; Behavioral: phone call
- 40 minute session, home practice e-health, no phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 40 minutes in duration. The daily home practice component for headache management will utilize a migraine specific interactive web portal, Migraine e-health portal. This arm will not receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 40 minute session; Behavioral: home practice e-health
- 40 minute session, home practice handout, phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 40 minutes in duration. The daily home practice component for headache management will utilize a handout with explanations of mind body skills and a home practice plan. This arm will also receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 40 minute session; Behavioral: home practice handout; Behavioral: phone call
- 40 minute session, home practice handout, no phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 40 minutes in duration. The daily home practice component for headache management will utilize a handout with explanations of mind body skills and a home practice plan. This arm will not receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 40 minute session; Behavioral: home practice handout
- 20 minute session, home practice e-health, phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 20 minutes in duration. The daily home practice component for headache management will utilize a migraine specific interactive web portal, Migraine e-health portal. This arm will also receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 20 minute session; Behavioral: home practice e-health; Behavioral: phone call
- 20 minute session, home practice e-health, no phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 20 minutes in duration. The daily home practice component for headache management will utilize a migraine specific interactive web portal, Migraine e-health portal. This arm will not receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 20 minute session; Behavioral: home practice e-health
- 20 minute session, home practice handout, phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 20 minutes in duration. The daily home practice component for headache management will utilize a handout with explanations of mind body skills and a home practice plan. This arm will also receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 20 minute session; Behavioral: home practice handout; Behavioral: phone call
- 20 minute session, home practice handout, no phone call (Experimental): This intervention arm consists of mind body skill introduction session that is 20 minutes in duration. The daily home practice component for headache management will utilize a handout with explanations of mind body skills and a home practice plan. This arm will not receive a follow up phone call 4 weeks after the introductory session to promote adherence to home practice.
  Interventions: Behavioral: 20 minute session; Behavioral: home practice handout

INTERVENTIONS:
Behavioral: 40 minute session — The 40 minute session will include all of the content contained in the 20 minute session, but will include a greater explanation of each of the mind and body skills, followed by in vivo practice of each skill with the nurse. Sessions will also include review of home practice for each group.
  Arms: 40 minute session, home practice e-health, no phone call; 40 minute session, home practice e-health, phone call; 40 minute session, home practice handout, no phone call; 40 minute session, home practice handout, phone call
Behavioral: 20 minute session — For participants randomized to the 20 minute session, content will include pain education, followed by brief explanations of each of the mind and body skills, in vivo diaphragmatic breathing practice and demonstration of use of biofeedback card. Sessions will also include review of home practice for each group.
  Arms: 20 minute session, home practice e-health, no phone call; 20 minute session, home practice e-health, phone call; 20 minute session, home practice handout, no phone call; 20 minute session, home practice handout, phone call
Behavioral: home practice e-health — Participants will be provided and instructed on access to a migraine-specific interactive web portal, Migraine e-Health. This web-based tool actively guides participants in practicing evidence-based mind and body skills. Use of the Migraine -e-Health application for the high dose capitalizes on teaching participants mind and body skills while increasing accessibility due to implementation on mobile devices.
  Arms: 20 minute session, home practice e-health, no phone call; 20 minute session, home practice e-health, phone call; 40 minute session, home practice e-health, no phone call; 40 minute session, home practice e-health, phone call
Behavioral: home practice handout — Participants will be given a handout of commercially available free apps relevant to the mind body skills introduced.
  Arms: 20 minute session, home practice handout, no phone call; 20 minute session, home practice handout, phone call; 40 minute session, home practice handout, no phone call; 40 minute session, home practice handout, phone call
Behavioral: phone call — The dose of phone call will occur about 4 weeks following the face-to-face mind and body introduction session and will last approximately 5-10 minutes. The phone call will be used to promote adherence to home-practice and answer questions related to skill use/home practice completion.
  Arms: 20 minute session, home practice e-health, phone call; 20 minute session, home practice handout, phone call; 40 minute session, home practice e-health, phone call; 40 minute session, home practice handout, phone call

SUMMARY:
This study uses a factorial research design to evaluate a nurse delivered mind body intervention using different doses of 3 treatment components to determine the optimized treatment for headache day reduction.

DETAILED DESCRIPTION:
In the United States, over 6 million children and adolescents suffer from migraine headaches and it is 1 of the 5 most prevalent childhood disorders. Mind and body approaches can significantly help these youth, but getting access to this type of treatment is a challenge for families. Our mind and body study will test a mind and body intervention package delivered by health care professionals (i.e., nurses) introducing coping skills to youth ages 10 to 17 that have migraine.

Using a factorial design and the multiphase optimization strategy "MOST", in this study we are able to evaluate different doses of 3 treatment components (1. Duration of mind and body skill introduction session; 2. Home practice support intensity; and 3. Adherence prompt phone call) in one project. A screening experiment will be conducted to determine the dose of each treatment component for future evaluation of the optimized intervention package in a pragmatic or SMART trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Migraine with or without aura or chronic migraine that meets the International Classification of Headache Disorders(ICHD) criteria
* Frequency: Headache frequency based upon prospective headache diary of 28 days must be ≥ 4 and ≤ 28.
* PedMIDAS: PedMIDAS Disability Score > 4, indicating at least mild disruption in daily activities and < 140, indicating extreme disability that may require more comprehensive, multi-component therapy
* Use of one or more of the following prescribed nutraceuticals and/or preventive anti-migraine medications at the time or randomization or be on a stable dose of one or more of the following throughout the 12 weeks of the study [Vitamin B2 (Riboflavin), Co-Q 10 (Coenzyme Q10), Magnesium (Mg), Vitamin D2 or D3 (Erocalciferol/Cholecalciferol), Depakote (Divalproate), Inderal (Propanerol), Elavil ((Amitripyline), Topamax (Topiramate), Periactin (Cyproheptadine)]
* Language: English speaking, able to complete interviews and questionnaires in English

Exclusion Criteria:

* Continuous migraine defined as unrelenting headache for a 28 day period
* Must agree not to take non-specific acute medication, such as NSAIDS (e.g., ibuprofen), more than 3 times per week, or migraine specific acute medications, such as triptans, more than 6 times per month (to prevent medication overuse headache)
* PedMIDAS Disability Score > 140, indicating extreme disability that may require more comprehensive, multi-component therapy
* Youth who are pregnant, or those who are sexually active and not using a medically accepted form of contraception (barrier or hormonal methods)
* Present severe psychiatric disease, alcohol or drug dependence, or documented developmental delays or impairments (e.g., autism, cerebral palsy, or mental retardation) or other circumstances, that, in the opinion of the investigator, would interfere with adherence to study requirements or safe participation in the study

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in number of headache days | baseline to post treatment (8 weeks post randomization)
  This outcomes measure examines whether the rate of absolute number of headache days, per 28 day period, differs between the treatment groups over time. This will be assessed longitudinally based on the actual number of headache days from the 28 days prior to randomization to the last 28 days before the endpoint visit.

SECONDARY OUTCOMES:
Change in absolute headache disability score on PedMIDAS | baseline to post treatment (8 weeks post randomization)
  The PedMIDAS scale which evaluates the impact of headaches in school, home, play, and social activities, is comprised of six items that pertain to days missed in various activities over the past 90 days. Questions are answered by the youth in consultation with their parents and reviewed by study staff. The PedMIDAS scale is administered at baseline (covering the three months prior to enrollment) and at the endpoint visit (covering three months of enrollment). A total PedMIDAS score (sum of items 1-6) was used in this study. Scores range from 0-240; with a score of 0-10 indicating no disability, 11-30 mild disability, 31-50 moderate disability, and more than 50 severe disability in daily activities.

OTHER OUTCOMES:
Feasibility and adherence to the session time component | baseline to post treatment (8 weeks post randomization)
  Thresholds will be used as guides to evaluate whether the assigned intervention is feasible and whether participants can adhere to that intervention. For the session time component a threshold of reasonable feasibility/adherence is specified as: nurse fidelity to introduction dose times (20 min versus 40 min) with fidelity measured as proportion of interactions where the documented time is within 5 minutes of the intended duration (i.e., 15 to 25 minutes for the 20-minute dose and 35 to 45 minutes for the 40-minute dose, as measured by nurse report at the time of the session). The acceptable threshold will be at least 80 percent fidelity within the given time window.
Feasibility and adherence to the home practice component | baseline to post treatment (8 weeks post randomization)
  Thresholds will be used as guides to evaluate whether the assigned intervention is feasible and whether participants can adhere to that intervention. For the home practice component a threshold of reasonable feasibility/adherence is specified as: eHealth versus handout - threshold >33% of practice days completed on average will be defined as sufficient adherence for both conditions.
Feasibility and adherence to the phone call component | baseline to post treatment (8 weeks post randomization)
  Thresholds will be used as guides to evaluate whether the assigned intervention is feasible and whether participants can adhere to that intervention. For the phone call component a threshold of reasonable feasibility/adherence is specified as: 50% of phone calls completed will be considered feasible/adherent for the phone call follow-up. No threshold is set for the participants who do not receive a phone call follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Powers, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - University of Colorado/Children's Hospital Colorado, Aurora, Colorado
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No